CLINICAL TRIAL: NCT06741956
Title: Design, Validation and Implementation of a Wearable Device for the Primary Prevention of Osteoporosis and Distal Radius Fractures in Women
Brief Title: Development of a Wearable Device for Osteoporosis Prevention and Fracture Risk Reduction in Women
Acronym: Weapom
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Collaborators: Hospitales Universitarios Virgen del Rocío (Other)
Responsible Party: Principal Investigator, Borja Sañudo, Head of the Department of Physical Education and Sport, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PID2022-142316OB-I00; PID2022-142316OB-I00 (Other Grant/Funding Number: Ministerio de Ciencia e Innovación)
Record Dates: First submitted 2024-12-10; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Osteoporosis in Post-menopausal Women; Prevention; Exercise; Physical Activity; Wearable Devices
Keywords: Osteoporosis prevention; Postmenopausal women; Bone mineral density; Fragility fractures; Physical activity interventions; Wearable technology; Non-pharmacological management; Machine learning in healthcare
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: The WEAPOM project is a single-blind (assessor), randomized-controlled trial. Eligible participants will be randomly assigned (1:1) to two groups: (i) a lifestyle modification program increasing impacts and physical activity level with a duration of 9 months (EV), or (ii) an unsupervised control group (CON) that will continue with their usual treatment.
Who Masked: Participant, Outcomes Assessor
Masking Description: The WEAPOM project is a single-blind, randomized-controlled trial where only the outcome assessors are blinded. Eligible participants are randomly allocated in a 1:1 ratio to one of two groups. The masking ensures that assessors evaluating outcomes are unaware of participant group assignments, reducing bias in the assessment of results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lifestyle intervention (Experimental): A. Program to increase physical activity and impacts For the intervention, a biosensor -wearable device- (Fitbit Versa) will be used. The device is linked to an App (Weapom) that will allow users to quantify the number of steps (including the rate of steps per minute), the impacts and their intensity. Users will be given feedback from the application on the level of achievement of the objectives proposed in the impact program (EV). It will be proposed to achieve 50 vertical and multidirectional jumps per day (milestone 1. The number of jumps> 3.9 G per day will be recorded 28, divided between 3-5 sets of 10-20 repetitions with a minimum 1-2 minute rest between sets. A frequency between 4-7 days per week will be used. In the same way, it will be recommended to reach 10,000 steps per day (milestone 2. The number of daily steps will be recorded) and, as far as possible, at a rapid pace (milestone 3. The number of daily minutes walking at a pace over 110 steps/minute will be
  Interventions: Behavioral: Weapom Lifestyle Intervention to measure bone impacts using a Fitbit Versa wearable device and the Weapom App.
- Control (No Intervention): Participants randomly assigned to CON will receive general advice from medical staff on the positive effects of physical activity and nutritional aspects for the prevention of osteoporosis. Participants in this group will carry the device, but will not have access to the App.

INTERVENTIONS:
Behavioral: Weapom Lifestyle Intervention to measure bone impacts using a Fitbit Versa wearable device and the Weapom App. — A. Program to increase physical activity and impacts For the intervention, a biosensor -wearable device- (Fitbit Versa) will be used. The device is linked to an App (Weapom) that will allow users to quantify the number of steps (including the rate of steps per minute), the impacts and their intensity. Users will be given feedback from the application on the level of achievement of the objectives proposed in the impact program (EV). It will be proposed to achieve 50 vertical and multidirectional jumps per day (milestone 1. The number of jumps> 3.9 G per day will be recorded 28, divided between 3-5 sets of 10-20 repetitions with a minimum 1-2 minute rest between sets. A frequency between 4-7 days per week will be used. In the same way, it will be recommended to reach 10,000 steps per day (milestone 2. The number of daily steps will be recorded) and, as far as possible, at a rapid pace (milestone 3. The number of daily minutes walking at a pace over 110 steps/minute will be r
  Arms: Lifestyle intervention

SUMMARY:
This project aims to determine the impact on bone health of:

A lifestyle intervention promoting impact-based activities and physical activity for nine months.

The same program enhanced with home-based strength training. A control group without supervision, continuing with standard care. The study will evaluate the persistence of changes after these interventions during a 12-week follow-up. By employing diverse strategies, the project seeks to identify barriers and facilitators to using technology for promoting healthy lifestyles in this demographic. Additionally, it will, for the first time in Spain, establish predictive models to assess the efficacy of non-pharmacological interventions in osteoporosis prevention, in collaboration with the public health system. These models will also predict adherence to technology-based behavioral interventions.

ELIGIBILITY CRITERIA

Eligible Participants:

Postmenopausal women aged >40 years, within 8 years post-menopause. Sedentary lifestyle. Willingness to provide informed consent.

Exclusion Criteria:

Surgically induced menopause or cancer treatment. Low BMI (<18 kg/m²). Excessive alcohol consumption (≥3 drinks/day). Smoking. Unstable cardiovascular disease, rheumatoid arthritis, chronic kidney disease. Diagnosed conditions altering bone metabolism (e.g., hyperthyroidism). Recent fractures or mobility limitations. Recent engagement in structured physical activity programs. Recent use of glucocorticoids or hormone replacement therapy. VARIABLES TO BE MONITORED Body Composition: Lean mass, fat mass, bone mass, and waist circumference. Bone Health: Bone density of lumbar vertebrae and femur via densitometry and microarchitecture evaluation using quantitative CT.

Biomarkers: Assessment of bone resorption and remodeling markers. Physical Function: Functional assessments (e.g., gait speed, jumping ability, lower limb strength).

Physical Activity: Objectively monitored with accelerometers, analyzing sedentary, light, and moderate-to-vigorous activities.

Nutritional Intake: Monitored using dietary recall tools. Quality of Life: Assessed using the Menopause Rating Scale (MRS). TRAINING PROTOCOL

A. Impact-Based Physical Activity Program:

Participants will utilize a validated biosensor (Muvone®) to track steps and impacts, targeting 50 multidirectional jumps and 10,000 steps per day, emphasizing brisk walking.

B. Home-Based Strength Training Program:

Two weekly sessions, progressing from 20 to 42 minutes, targeting major muscle groups (e.g., squats, hip extensions). Sessions include warm-ups, multi-joint exercises, and recovery periods.

C. Control Group:

Participants receive general advice on physical activity and nutrition without supervised programs or app access.

FOLLOW-UP After 36 weeks, participants will resume daily routines without app feedback. At the 12-week follow-up, they will return for questionnaires and physical assessments.

This structured approach ensures rigorous evaluation and facilitates integration of findings into public health strategies.

DETAILED DESCRIPTION:
CURRENT STATUS AND JUSTIFICATION OF THE PROPOSAL Osteoporosis is an important public health problem and it is characterized by the deterioration of the microarchitecture of bone tissue and a low bone mineral density (BMD) that leads to a reduction in bone strength and the consequent increased risk of skeletal fractures 1. One in three women will suffer an osteoporotic fracture in their lifetime 2. In fact, it is estimated that more than 200 million people suffer from osteoporosis and these figures are increasing due to the aging of the population and the change in lifestyles 3. A recent systematic review gathered epidemiological information on selected musculoskeletal injuries and provided pooled injury-specific incidence rates. Authors reported that the most common fractures in the whole adult population based on the pooled incidence rates were distal radius fractures (212 per 100,000 person-years)4. Distal radius fractures account for one in five bony injuries in both primary and secondary care5. According to data from the International Osteoporosis Foundation (IOF), in Spain there would be more than 2.8 million women over the age of 50 with osteoporosis, with more than 330,000 fragility fractures per year and projections suggest that by 2030 these figures will increase 28.8%1. Consequently, there is a significant economic burden on the healthcare system for patients who experience an osteoporosis-related fracture. Direct costs for osteoporosis, such as medications, occupational therapies, and inpatient and outpatient visits, are expected to increase to $25 billion by 2025 as the population ages 6. Together with the indirect costs, such as loss of productivity, are expected to rise to more than $95 billion in 2040 6. Osteoporosis, and the 4.3 million fragility fractures that it causes, cost the health care systems of Europe over €56 billion each year based on data for 2019 7. Only in our country it is estimated that the cost associated with sick days due to fragility fractures amounts to €355,000 each year. Only the direct and indirect costs associated with these fractures would exceed €4.2 billion, with a projected increase of 30.6% by 2030 1. It should not surprise us, therefore, that in postmenopausal women, osteoporotic fracture costs exceed the annual costs for breast cancer, myocardial infarction (MI), and stroke 6.

The loss of the protective effect of estrogens on the skeletal structure after menopause intensifies the decrease in bone density as a result of a sudden imbalance between bone formation and bone resorption. This decrease in estrogens (e.g., estradiol) leads to an increase in the rate of bone remodeling due to an increase in the number of osteoblasts and osteoclasts; although osteoclast-mediated removal of bone matrix is much greater than osteoblast bone formation8. Therefore, the loss of BMD is very evident, especially in the 3-5 years following the last menstrual period 9, in a 2% loss rate per year 10. Parallel to this decrease in BMD, it is common to find a decrease in muscle mass and strength, probably derived from the decrease during menopause of certain precursors (e.g., insulin-like growth factor type 1, -IGF-1-) 11. It is important to note that bone strength is determined not only by bone mass, but also by the size, shape, structure, or properties of collagen 12. Since densitometry (DEXA) captures only bone mass, there is growing interest in the use of other three-dimensional imaging modalities, such as quantitative computed tomography (QCT) to assess bone strength. QCT can help differentiate between the cortical and trabecular compartments of bone and their relative contribution to bone strength in vivo. Similarly, various biomarkers have been identified to detect the dynamics of bone remodeling 13,14. The National Bone Health Alliance and the American Association for Clinical Chemistry have suggested that the most widely accepted biomarkers for the evaluation of interventions in osteoporosis are the C-terminal telopeptide of collagen type 1 -CTX-1- (bone resorption) and the amino-terminal propeptide of procollagen type 1 -P1NP- (bone formation) 13,14.

There are well-known modifiable and non-modifiable risk factors for osteoporosis. Non-modifiable items would include age, family history of fragility fractures, type 1 diabetes, rheumatoid arthritis, or cancer treatment (e.g., aromatase inhibitors or chemotherapy). In the first group, smoking, excessive alcohol consumption, the use of corticosteroids, insufficient calcium or vitamin D, low body mass index (BMI), sedentary lifestyle15, or the lack of physical activity, which would be another of the main risk factors can be included. However, bone loss can remain clinically silent. A recent retrospective healthcare study found that 79.4% of patients did not have a diagnosis or treatment on-board for osteoporosis 12 months before the fracture 6. It surprises that less than half of women at high risk of fracture are treated despite the high cost of fractures and the availability of affordable medications 2. Consequently, according to the IOF, there is a large unmet need as it relates to the prevention of postmenopausal osteoporosis because many women are not undergoing the recommended diagnostic screenings or assessing baseline osteoporosis risk 15.

Prevention should be the priority when pursuing the reduction of the burden caused by osteoporosis16. In addition to prevention, the optimization of the management, from first aid to rehabilitation, should be well considered to reduce excess costs. The approach in this population group is usually multimodal and includes both pharmacological and non-pharmacological interventions. In Europe, the most commonly used drugs for osteoporosis are bisphosphonates, raloxifene, parathyroid hormone drugs, and denosumab 17. However, the widespread and long-term use of these drugs is limited due to possible side effects 18. Therefore, diet and physical exercise, together with other environmental and lifestyle factors, would constitute the main non-pharmacological strategies for the management of this pathology 19. However, although physical activity is a modifiable factor that contributes to the improvement of bone mass and strength, our understanding of how to quantify the dimensions of physical activity that are osteogenic (including frequency, intensity, time, and type) is incomplete. There is no doubt that to initiate an osteogenic response, the bone must be subjected to a stimulus that exceeds a threshold determined by the usual range of deformation in the predominant load direction19. Precisely, the mechanical stress to which exercise (impacts and muscle contraction) subjects the bone (e.g. tension, compression, hydrostatic pressure) can promote osteogenic differentiation of mesenchymal stem cells, increasing osteoblastic regulation through different mechanisms 20. To increase effectiveness, the exercise must: (i) be dynamic, not static; (ii) exceeding an intensity threshold; (iii) exceeding a strain frequency threshold; (iv) be relatively short but intermittent; (v) imposing an unusual load pattern on the bones; (vi) include adequate availability of calcium and vitamin D 21. However, the optimum loading patterns of bone that produce clinically significant benefits have not been clearly defined to date, since it has not been possible to easily quantify exercise intensity in terms of bone-loading forces in clinical settings22. Q1

Recent guidelines for the prevention and management of osteoporosis through physical exercise suggest interventions that last longer than 8 months and that combine high impacts and high-intensity strength training. Interventions in which fast walking (e.g., > 6 km/h) is combined with activities that incorporate a relatively short number of impacts (e.g., 10-50 jumps per day), at intensities exceeding 2-4 times body weight (~ 3.9 G), at least 4 sessions a week and using multiaxial exercises to generate an unusual load on the hip, can help postmenopausal women to compensate for age-related bone loss 23. These would be effective strategies to preserve BMD in postmenopausal women with a level of evidence 1a24. However, there is no evidence of its effectiveness in preventing distal radius fractures Q2 and also dropout rates in these types of programs are high25 and, despite the evidence, participants are often reluctant to exercise, citing barriers as poor health, lack of time due to family responsibilities, lack of companionship or encouragement, lack of access to adequate facilities or opportunities, or cost. Patients with osteoporosis often report a lack of time and transportation limitations as the main barriers that would limit their participation in supervised training programs 26. For these reasons, it has been suggested that intervention trials should use settings that are easily accessible to participants and provide flexible exercise schedules 25.

In the literature, it is suggested that in interventions aimed at bone health in young adult women, it is crucial to minimize the perceived demands of time (e.g., short and flexible intervals) and environmental barriers related to the convenience and accessibility of physical activity 25. Therefore, to increase adherence in this population group, regular contact with study personnel, personalization of progression, and adequate exercise monitoring (avoid safety concerns and lack of confidence) are suggested. In a recent study from our group, evidence showing that non-supervised exercise programs could be effective to improve BMD in adult women was found. However, only five studies were available in postmenopausal women and overall registered a substantial dropout rate (above 40%) due to unwillingness to continue and illness among the main reasons. Therefore, the necessity to investigate the efficacy of remote/assistive technologies for delivering and monitoring non-supervised exercise interventions was highlighted. The question that should be asked is, in what way all these issues can be managed, facilitating the monitoring of the program and solving the barriers outlined?

Mobile and digital technologies (mHealth) allow complementing exercise programming for the management of osteoporosis by providing information on skeletal mechanics during locomotion23. However, and even though wearable activity trackers offer potential as a multifaceted intervention to help people become more active, no study has examined the usefulness of these wearable devices in postmenopausal women nor in the upper extremities Q3. The importance of reaching a minimum threshold of stimulation to obtain bone adaptations has been justified, since insufficient loads would not have the desired effect, for this reason, precise quantification of the mechanical loads to which the musculoskeletal system is subjected is necessary, what could be achieved with certain biosensors28. However, interventions based on this type of technology aimed at preventing osteoporosis are very scarce29, even though authors agree on their potential, not only for increase the benefits of the interventions, but mainly to improve adherence to them.

In summary, the scientific community face a group of women with a high risk of suffering from osteoporosis (potential incidence of fragility fracture), with the subsequent incidence for their functionality and quality of life, on the one hand, and for the health system, on the other. The strategies for managing this group suggest the incorporation of activities that require impact and strength training; however, direct measurement of bone strains requires invasive surgical procedures and indirect measurement of ground reaction forces are limited to a fixed place and time, being thus impracticable in long-term clinical measurements. Assessing the effects of this type of intervention could help to record variables that, after proper analysis (e.g., machine learning), facilitate decision-making and reduce the use of resources in the health system. Therefore, the questions that arise are: ¿can indirect surrogate of bone strains that are now readily measurable with a novel accelerometer-based measurement device be used? ¿Can these wearable devices be used to investigate the effect of exercise-induced impact loading on bone mineral density, geometry and metabolism in posmenopausal women with the intention of assessing the intensity and amount of impact loading required to gain adaptive effects at the wrist level? Starting hypothesis: The lifestyle intervention controlling the intensity of impact and exercises with wearable devices will improve bone composition and structure, physical fitness and quality of life in postmenopausal women. Evaluating the effect of a bone-targeted exercise training programme on extra-skeletal risk factors of osteoporotic fractures and physical performance scientist will be able to design a technological smart cloud platform with digital technologies (artificial intelligence, a mobile-based application and wearable managed in the cloud) that could be implemented (after the proper identification key factors for the transfer of research results obtained in the experimental phase) to the public socio-health system contribute in the prevention of osteoporosis and frailty fractures.

Procedures

Objective 1 Participants will be scheduled for three days to complete the measurement protocol. On the first day, they will attend the hospital and complete the sociodemographic and clinical information. They will then receive the accelerometer and all the questionnaires to be completed at home. In addition, from the hospital center, the participants will be cited another day for the biochemical analysis, QCT and densitometry. On a second day, the participants will be cited to the university laboratory to return the accelerometers and questionnaires, and they will take the physical fitness tests. Finally, in a third visit to the laboratory, the participants will be familiarized with the use of the recording wearable. Finally, all participants will receive a daily vitamin D supplement of 600 IU/day. If serum levels are deficient, it will be supplied for 4 months: 1 vial of 25,000 IU per month if <20ng/ml, 1 vial of 25000 IU every 15 days if <15ng/ml, 1 vial of 25,000 IU every week if <10 ng/ml. Calcium intake will be calculated using the 3-day recall and supplemented up to 1200 mg per day.

Lifestyle intervention

A. Program to increase physical activity and impacts For the intervention, a biosensor -wearable device- (Fitbit Versa) will be used. The device is linked to an App (Weapom) that will allow users to quantify the number of steps (including the rate of steps per minute), the impacts and their intensity. Users will be given feedback from the application on the level of achievement of the objectives proposed in the impact program (EV). It will be proposed to achieve 50 vertical and multidirectional jumps per day (milestone 1. The number of jumps> 3.9 G per day will be recorded 28, divided between 3-5 sets of 10-20 repetitions with a minimum 1-2 minute rest between sets. A frequency between 4-7 days per week will be used. In the same way, it will be recommended to reach 10,000 steps per day (milestone 2. The number of daily steps will be recorded) and, as far as possible, at a rapid pace (milestone 3. The number of daily minutes walking at a pace over 110 steps/minute will be recorded, as this is considered the threshold of moderate-vigorous intensity in this age range 40. Therefore, according to the new WHO guidelines 41 on physical activity and sedentary behavior, it will be quantified whether 150 minutes a week of moderate-vigorous physical activity are achieved. In addition, and in order to specifically focused on radius strength, 50 (3 to 5 cm) drops with the arms completely straight will be register. In parallel, the participants in both groups will receive recipes rich in calcium through the App and will have a calculator to calculate the intake of calcium and other micronutrients through the diet. They will also receive information on osteoporosis and strategies for its prevention (e.g., advice on sun exposure).

B. Control group Participants randomly assigned to CON will receive general advice from medical staff on the positive effects of physical activity and nutritional aspects for the prevention of osteoporosis. Participants in this group will carry the device, but will not have access to the Muvone App.

Objective 2 Upon placement of the accelerometers, participants completed a standardized exercise protocol during a laboratory-based activity session. The exercise protocol consisted of five countermovement jumps (CMJ) with a 30 s rest between each jump. The jump height was measured with a light barrier system (OptoGait, Microgate, Bolzano, Italy). Participants then performed four treadmill activities (HP-Cosmos®, Traunstein, Germany), walking/running at 4.8, 6.4, 9.7 and 12 km·h-1.The duration of each treadmill bout was 2 min with a 1 min rest between each condition. Participants stood still during rest intervals and completed every exercise protocol in a randomized order. To evaluate spatio-temporal gait parameters during the protocol, a floor-based photocell system (OptoGait, Microgate, Bolzano, Italy) was used. Finally, participants will be instructed to fix their shins on a soft pillow and extend their knees to lean forward. The thigh will be set at 30º from the horizontal. Participants will be raised to reach a proper height from the ground (3 cm or 5 cm between the palm of the hand and the force plates). The subjects will be instructed to keep their elbows fully extended (i.e. outstretched hands) and the arm angle will be set at 15° to the vertical. Each participant will complete ten trials, which involved five trials at h=3 cm, 15 minutes of rest, and five experiments at h=5 cm.

To assess the intensity and amount of impact loading, the vertical acceleration peak values will be recorded with an accelerometer based human body movement monitor (Fitbit). The monitor was worn on a wrist 2 cm above the medial epicondyle. For the individual quantification of their daily physical activity, all participants will be asked to carry the monitor during all waking hours for 36 weeks. The number of daily acceleration peaks will be recorded at 33 acceleration levels from 0.3 to 9.9 g. The individual daily average number of peaks at each acceleration level will be calculated for the analysis. The number at different acceleration levels will be analysed to describe the intensity of exercise. Previously, the reliability of the accelerometer-based method using a three-dimensional prototype was tested. However, in this project, the impacts at the wrist level will be measured. The peak values were predominantly obtained immediately after heel contact in different activities; furthermore, the peak acceleration values will be compared with the values obtained simultaneously using a standard optical motion analysis system. Moreover, the acceleration values will also be compared with the GRF measured with a force plate (Kistler 9287A, Kistler Instrument, Switzerland), with the acceleration values multiplied by body weight.

Objective 3 In order to identify the key factors for the transfer of research results obtained in the experimental phase to the public socio-health system, the results will be discussed in 3 meetings by a group of experts in the health system (e.g., a district director of Primary Care centers or a politician from the health area of the Junta de Andalucía, two directors of primary care centers, an expert in health promotion, a nurse in care of patients with osteoporosis, etc.). Different models will be designed using biochemical, image, clinical and physical condition data that guide medical personnel on the most relevant factors that determine the response to this type of treatment. Out the whole set of variables included on the electronic healthcare records, a new medical model including only the selected high impact variables (sub-dataset) calculated with machine learning feature selection techniques will be designed. The health gain (QUALYs) and costs will be determined, and the cost-effectiveness ratio (ICUR) will also be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women older than 40 years with ≤ 10 years after menopause ("early postmenopausal women").
* Sedentary women (defined as not performing regular physical activity greater than 150 min of moderate-vigorous physical activity per week in the last six months).
* Willing to give consent to participate in the study.

Exclusion Criteria:

* Surgically induced menopause or cancer treatment.
* Low BMI (<18 kg / m2).
* Excessive alcohol consumption (≥3 drinks per day).
* Smoker
* Unstable cardiovascular disease.
* Rheumatoid arthritis.
* Chronic kidney disease
* Diagnosis of conditions that alter bone metabolism (hypo/hypercalcemia, hyperthyroidism, hypo/hypergonadism).
* Upper or lower limb fracture in the last 6 months.
* Mobility problems or requiring assistance to walk.
* Participation in physical exercise programs in the 6 months prior to the study.
* Regular use of glucocorticoids or hormone replacement therapy in the past 3 months.
* Unwillingness to complete the study requirements.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The eligibility for this study is based on biological sex due to the specific focus on postmenopausal osteoporosis, a condition influenced by physiological and hormonal changes that occur in women after menopause. Gender identity does not limit participation, provided the individual meets the inclusion criteria based on biological and physiological factors associated with postmenopausal status.
Enrollment: 120 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Bone density | Pre (week 0) and post (week 36).
  The BMD (g/cm2) of the lumbar vertebrae (L1-L4) and femur of the right leg (femoral neck, Ward's triangle, and greater trochanter) will be analyzed by a specialist technician outside the study. Values will be converted to T-score and Z-score based on the reference values for a Caucasian female and the bone density of the Spanish population, respectively. The device will be calibrated daily using a phantom.
Bone biomarkers | Pre (week 0) and post (week 36).
  To avoid diurnal variation, fasting blood samples will be collected between 8:00 and 10:00 in vacutainer tubes and aliquots will be stored frozen at -80ºC until analysis. Serum Β-CrossLaps (β-CTX) to assess bone resorption and P1NP, to assess bone remodeling, will be measured both at baseline and at 36 weeks by chemiluminescence (ECLIA) on a Modular Analytics E170 analyzer (Roche Diagnostics, Switzerland).

SECONDARY OUTCOMES:
Body composition | Pre (week 0) and post (week 36).
  Whole-body lean, fat, and bone mass will be measured using a DEXA device (Hologic Horizon Wi, Waltham, MA, USA). Lean Mass: Reported in kilograms (kg), representing the total body weight minus fat and bone mass.
  Fat Mass: Expressed in kilograms (kg) and as a percentage of total body weight (%).
Quality of life | Pre (week 0) and post (week 36).
  The quality of life of the participants will be determined with the Short-Form Health Survey 36 (SF-36). The SF-36 is a generic instrument to assess health-related quality of life. It contains 36 items grouped into 8 dimensions: physical functioning, physical role, body pain, general health, vitality, social functioning, emotional role and mental health. The score ranges from 0 to 100 in each dimension, with higher values indicating better health.
Symptoms of menopause | Pre (week 0) and post (week 36).
  Participants will complete the Menopause Rating Scale (MRS) questionnaire, which is a menopause-specific quality of life scale developed and validated to assess the severity of symptoms related to menopause. It consists of 11 items, which cover three dimensions: (1) somatic symptoms, which include vasomotor symptoms, cardiac discomfort, sleep problems, and joint or muscle discomfort (items 1-3 and 11, respectively); (2) psychological symptoms, including depressed mood, irritability, anxiety, and physical or mental exhaustion (items 4 to 7, respectively); and (3) urogenital symptoms, including sexual problems, bladder problems, and vaginal dryness (points 8 to 10, respectively). A five-point rating scale for each item allows participants to describe the perceived severity of symptoms (no complaints, 0; mild, 1; moderate, 2; severe, 3; and extremely severe, 4). The subscales are analyzed by summing the individual scores for each subscale. A value of 17 is used as a cut-off point to d
Mobility and dynamic balance | Pre (week 0) and post (week 36).
  Timed up and go (TUG), which consists of getting up from a chair without using your hands, walking a distance of 2.44 m, turning around a cone and sitting down again. Two trials will be carried out with 3 min rest between them, registering the best time (in seconds).
Strength | Pre (week 0) and post (week 36).
  To estimate strength and power gains in response to the training program, isometric strength (90 ° flexion at the knee and 20 ° at the hip) and isokinetic strength in concentric (at angular velocities of 60 and 240°s- 1) and eccentric (120 °·s-1) in flexion and extension of the knee and hip, using an isokinetic dynamometer (Biodex System 4; NY, USA). The peak of the torque and the average power of each series will be recorded
Jump ability | Pre (week 0) and post (week 36).
  The maximum impulse (N s) of the vertical reaction forces against the ground in a vertical countermovement jump (CMJ) on a platform will be evaluated. force (Kistler, Winterthur, Switzerland). Participants will perform 3 CMJ with 1 min rest between them, registering the best value for future analyzes.
Physical activity and sedentary behavior | Pre (week 0) and post (week 36).
  Accelerometry will be used to objectively evaluate physical activity and sedentary time. Participants will be asked to use a wearable accelerometer for 9 consecutive days, beginning on the same day they receive the monitor (e.g., participants who receive the accelerometer on Monday, will carry the device until Tuesday of the following week). The first and last days will be excluded from the analyzes, accounting for a total of 7 days of registration. Participants will be instructed to wear the accelerometer throughout the day (24 h) on the non-dominant hip. They can only remove it to shower, practice water sports and sleep. Only the data of those accelerometers that record at least 4 days with a minimum of 10 hours of recording will be included. The data will be filtered and transformed into counts per minute (CPM). Sedentary, light and moderate to vigorous physical activity time (MVPA).
Eating patterns | Pre (week 0) and post (week 36).
  The Mediterranean Diet Score, created to evaluate the degree of adherence to the traditional Mediterranean dietary pattern. It consists of 11 items (unrefined cereals, potatoes, fruits, vegetables, legumes, fish, olive oil, red meat and derivatives, poultry, dairy products and alcohol), whose scores range from 0 to 5 depending on the frequency of consumption.
Adherence to the program and adverse effects | Pre (week 0), week 20 and post (week 36).
  Compliance with the home exercise program will be recorded in training diaries. Before each training session, participants will rate muscle pain on a 10-point visual analog scale (min 0 - max 10); any fall or fracture; and any changes in physical activity, diet, or medications since the last training session will be recorded in the training diary.
Health gain and costs | Pre (week 0) and post (week 36).
  Health gain will be determined in quality-adjusted life years (QALYs), whereas, for costs, a health system perspective will be used, and the outputs were the difference in total health system costs between business-as-usual and the modeled intervention and included the cost of implementing the intervention. The incremental cost-effectiveness ratio (ICUR) will be calculated as the incremental cost of the intervention divided by the difference in QALYs between the groups. The 95% confidence interval of incremental QALYs between groups and ICUR will be calculated using non-parametric bootstrapping technique and plotted a cost-effectiveness acceptability curve with the main aim of calculating the probability that the intervention is cost effective. We will also calibrate the model for other epidemiological aspects included in the outcomes (e.g., age, medication or function).
Waist circumference (cm) | Pre (week 0) and post (week 36).
  Waist circumference (cm) will be assessed midway between the ribs and the crest of the ileum, with the participant standing (Harpenden tape, Holtain Ltd).
Height | Pre (week 0) and post (week 36).
  A stadiometer (SECA, Hamburg, Germany) will be used to measure the height (in cm) of the subjects without shoes.
Lower-limb strength | Pre (week 0) and post (week 36).
  The 30 s chair stand test (30 s-CST), in which the number of times in 30 s that the participant can get up from a chair to stand fully from a sitting position with a straight back and feet supported is counted on the ground, without leaning on the arms.
Walking speed | Pre (week 0) and post (week 36).
  To assess the speed of the walk, the participants will walk as fast as possible a distance of 5 m. The speed (m·s-1) will be evaluated using a photocell system (Racetime 2; Microgate, Bolzano, Italy).
Food frequency | Pre (week 0) and post (week 36).
  A food frequency questionnaire (FFQ) will be used that will allow a detailed description of the type and quantity of food and beverages consumed during 3 consecutive days (two ordinary days and one weekend).

CONTACTS AND LOCATIONS:
Overall Officials: Borja Sañudo, PhD, Principal Investigator — University of Seville; Sergio Tejero, PhD, Principal Investigator — Hospitales Universitarios Virgen del Rocío
Locations (1):
- Hospital Universitario Virgen del Rocío, Seville, Spain, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Once processing, quality control, analysis and publication are complete, the data will be made accessible in open access repositories. These data will be anonymized (remove potentially identifying information).

REFERENCES:
- [Derived] Sanudo B, Reverte-Pagola G, Maher C, Godino J, Carrasco L, Oviedo MA, Feria A, Sanchez-Trigo H, Gamboa H, Domingo-Molina R, Sanchez-Arteaga A, Giraldez MA, Martinez-Maestre MA, Cepeda E, Ladron-de-Guevara C, Rangel C, Pecci J, Farrahi V, Tejero S. Effectiveness of an mHealth-based impact exercise program for bone health in postmenopausal women: a randomised controlled trial protocol. BMC Public Health. 2025 Jul 10;25(1):2426. doi: 10.1186/s12889-025-22576-9. PMID 40640761